CLINICAL TRIAL: NCT01463436
Title: Study of Soy Isoflavone 100 mg/Day in Postmenopausal Women to Elaborate the Effect of Soy Isoflavone in Endothelial Function and to Reduce Oxidative Stress
Brief Title: The Effect of Soy Isoflavone Supplementation on Endothelial Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trisakti University (Other)
Responsible Party: Principal Investigator, Dr. dr. Pusparini SpPK, Principal investigator, staff of Clinical Pathology Department, Trisakti University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Usakti
Record Dates: First submitted 2011-10-25; First posted 2011-11-01 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Cardiovascular Disease; Osteoporosis
Keywords: endothelial function; postmenopausal; soy isoflavone supplementation; osteoporosis
MeSH Terms: conditions — Cardiovascular Diseases; Osteoporosis | interventions — Soybean Proteins; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- soy isoflavone 100 mg (Experimental): the experimental group receiving tablet contain soy isoflavone 100 mg and calcium carbonate 500 mg
  Interventions: Dietary Supplement: soy isoflavone
- calcium carbonate 500 mg (Placebo Comparator): The control group receiving a tablet contains calcium carbonate 500 mg for 6 months and 12 months
  Interventions: Dietary Supplement: control group

INTERVENTIONS:
Dietary Supplement: soy isoflavone — 100 mg soy isoflavone tablet containing genistein 55%, daidzein 39% and glycitein 6% and calcium carbonate 500 mg in the experimental group for 6 months and 12 months
  Other Names: kacang kedelai, soya bean
  Arms: soy isoflavone 100 mg
Dietary Supplement: control group — the control group receiving tablet contain calcium carbonate 500 mg/day for 6 months and 12 months
  Other Names: plasebo
  Arms: calcium carbonate 500 mg

SUMMARY:
A randomized double blind controlled trial was conducted to evaluate the effect of daily supplementation with soy isoflavone 100 mg/day for 12 months on 182 postmenopausal women aged 47 to 60 years at subdistrict South Jakarta Indonesia. The study hypothesis was supplementation soy isoflavone 100 mg/day for 6 and 12 months can increase endothelial function.

DETAILED DESCRIPTION:
The subject were randomized to the intervention group receiving tablets consisting of 100 mg soy isoflavone and calcium carbonate 500 mg and the control group receiving 500 mg calcium carbonate for 1 year. This study was carried out 13 months(13 x 28 days).

There were three outcome measure from this study; vascular cell adhesion molecule-(VCAM-1), nitric oxide (NO) and malonyldialdehyde (MDA). The outcome measure will be assessed at three times; before soy isoflavone supplementation / the beginning of study,post supplementation 6 months and 12 months. The outcome will be measured change from baseline in the level of VCAM-1, NO and MDA.

ELIGIBILITY:
Inclusion Criteria:

* healthy postmenopausal women
* natural cessation 1-10 years
* body mass index <=35 kg/m2
* not receiving medication and supplement in the previous 6 months

Exclusion Criteria:

* has chronic or terminal disease
* severe psychosis

Ages: 47 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
the changes levels of endothelial function marker in blood after 13 months supplementation | 13 months
  this study were measured the change levels of vascular cell adhesion molecule-1 (VCAM-1), nitric oxide (NO) as endothelial function parameter and malonyldialdehide as lipid peroxidation parameter from baseline to 6 months supplementation and from baseline to 13 months supplementation

SECONDARY OUTCOMES:
the changes levels of osteoporosis parameter after 6 months supplementation | 6 months
  This study have another outcome such as rank ligand, C telopeptide and osteoprotegrin as marker of osteoporosis. We will be measured the changes levels of osteoporosis marker after 6 months supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Pusparini Sunarno, Doctor, Principal Investigator — Trisakti University
Locations (1):
- Trisakti University, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Hall WL, Rimbach G, Williams CM. isoflavones and endothelial function. Nutrion Research Review 18:123-131, 2005. Vincent A,Fitzpatrick LA. soy Isoflavone: are they useful in menopause? Mayo clinic Proceeding 75:1171-1184, 2000
- See also: click here for more information about this tudy — http://www.univmed.org